CLINICAL TRIAL: NCT00627991
Title: The Use of Valsartan for the Management of Blood Pressure in Acute Stroke: Effects on Cerebral Blood Flow.
Brief Title: Blood Pressure Lowering in Acute Stroke Trial (BLAST)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Gregory W Albers, Principle Investigator, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SU-01282008-990; 7599
Record Dates: First submitted 2008-02-22; First posted 2008-03-04 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke | interventions — Valsartan

INTERVENTIONS:
Drug: Valsartan

SUMMARY:
Patients who are suffering from a stroke often present to the hospital with elevated blood pressure. Elevated blood pressure in the setting of stroke increases the risk of brain swelling or bleeding into the brain. Even so, there has been concern about lowering the blood pressure with medications because the newly injured parts of the brain may not get the blood flow they need, thereby worsening the damage from the initial stroke. We hope to demonstrate that the drug valsartan can be used safely and modestly to lower blood pressure in acute stroke patients, without having a detrimental effect on brain blood flow or neurologic status. Novel MRI techniques to measure brain blood flow will be used in conjunction with clinical scales to demonstrate safety.

DETAILED DESCRIPTION:
Hypertension is an important modifiable risk factor for the prevention of ischemic stroke. Whether specific antihypertensive medications confer an added benefit for recurrent stroke reduction beyond their ability to lower blood pressure remains a controversial subject. Because of their varied mechanisms of action, and their potential role as neuroprotective agents, there has been particular interest in drugs that affect the renin-angiotensin-aldosterone system (RAAS). Several large multi-national randomized clinical trials have suggested a unique benefit of these agents, namely angiotensin converting enzyme (ACE) inhibitors and ARBs, for the prevention of vascular events. Even with the very modest reductions in blood pressure achieved in the HOPE trial, ramipril was found to have a significant benefit on recurrent stroke prevention (Heart Outcomes Prevention Evaluation Study Investigators, 2000). In the LIFE study, losartan was shown to be more efficacious for the prevention of recurrent strokes in hypertensive patients than atenolol, despite nearly identical reductions in blood pressure (Dahlöf et al, 2002). This is an area of some debate, however, as some data may support the lowering of blood pressure in general over the use of specific agents such as ACE inhibitors for the prevention of recurrent stroke (PROGRESS Collaborative Group, 2001). More recently, the ACCESS study showed a benefit of early treatment with candesartan cilexetil on 12-month mortality and the number of vascular events in patients who had suffered an acute stroke (Schrader et al, 2003). The mechanisms that underlie this are uncertain, but the study suggests that early treatment of blood pressure in acute stroke may have long-term benefits, presumably independent of hemodynamic factors.

The use of antihypertensives in the setting of an acute infarct is an area of great interest. A transient rise in blood pressure is frequently seen in acute stroke patients (Semplicini et al, 2003). Although blood pressure typically normalizes within one week without treatment, about one-third of patients remain hypertensive (Britton et al, 1986; Harper et al, 1994). Currently, there is insufficient data for a clear recommendation on deliberately altering blood pressure in these acute ischemic stroke patients (BASC, 2004). That being said, hypertension in acute stroke has been associated with poor outcome (Warlow et al, 1996), although the relationship may be a 'J'-shaped curve, with both low and high mean blood pressures being detrimental (Leonardi-Bee et al, 2002). The potential mechanisms that underlie the association between hypertension and poor outcome in acute stroke are several, but may include an increase in peri-infarct edema and an increased risk of hemorrhagic transformation. The potential benefits of the early treatment of high blood pressure in acute stroke must be weighed against the theoretical risk of worsening ischemia in compromised neural tissue. The INWEST trial showed increased mortality in patients actively treated with a calcium-channel blocker within 72 hours of an acute stroke (Wahlgren et al, 1994), an effect that may be related to the lowering of diastolic blood pressure (Ahmed et al, 2000). This data is in keeping with the long-standing hypothesis that impaired autoregulation in the ischemic brain tissue renders cerebral blood flow purely pressure-dependent. A decrease in systemic blood pressure would then translate to decreased local perfusion to vulnerable tissue in the ischemic penumbra. It is in this setting that drugs that modulate the RAAS may have a unique role. In recent years, animal and human data has accrued that suggests CBF is maintained with these agents, even in the face of decreased systemic blood pressure.

There are human data regarding cerebral blood flow and drugs that affect the RAAS, in both normal patients and those with recent ischemia. Studies with ACE inhibitors have demonstrated a moderate lowering of blood pressure in hypertensive patients, without a corresponding decrease in CBP, as measure with xenon CT (Minematsu et al, 1987; Waldemar et al, 1990). Dyker et al (1997) used Doppler ultrasound to show that cerebral blood flow is maintained in the setting of acute stroke when systemic blood pressure is lowered with perindopril. A similar result was seen in hypertensive stroke patients with moderate to severe internal carotid artery stenosis or occlusion (Walters et al, 2001). When losartan was introduced in hypertensive patients within 2-7 days of a mild ischemic stroke, there was no adverse effect on global or region cerebral blood flow, as measured by carotid Doppler and brain hexamethylpropyleneamine oxime single photon emission computed tomography (HMPAO SPECT; Nazir et al, 2004). There is no published data on the effects of these drugs on cerebral perfusion as measured with MRI, nor on changes in infarct volume as measure by DWI.

Brain imaging with MRI is available at all major centers that admit patients for the care of ischemic stroke. Diffusion-weighted imaging is considered the 'gold standard' for the detection of ischemia in the acute setting, with restricted diffusion being visible within 30 minutes of symptom onset (Fisher and Albers, 1999). Semi-quantitative measures of cerebral blood flow can be obtained with perfusion-weighted imaging (PWI) with only a minimal increase in the total scanning time. The acquisition of perfusion data with MRI is more readily available than such modalities as PET, SPECT, or xenon CT. Data is ongoing to identify analysis regimens for PWI that best represent true cerebral perfusion. We will use these techniques to assess brain perfusion before and after the lowering of blood pressure with valsartan.

We hope to show that valsartan can be used safely in the setting of acute stroke to lower elevated blood pressure. There are novel properties of this class of drug (an angiotensive-receptor blocker or ARB), and promising human and animal data, that would suggest this drug can be safely used to lower blood pressure in the setting of acute stroke without compromising brain blood flow (i.e. cerebral perfusion). If this is proved to be the case, this compound could potentially be used routinely in this setting, with the hope of improving outcome. This pilot study may pave the way for a larger randomized trial looking at outcome measures in stroke patients. Further, a positive result in the this pilot study will serve as proof of concept that ARBs maintain cerebral perfusion while decreasing blood pressure, an overall favorable property.

ELIGIBILITY:
Inclusion Criteria:

1. Men and non-pregnant women over age 18 who have had an acute ischemic stroke referable to the anterior circulation, as diagnosed by one of more of the following: clinical judgment, head CT, and/or MR imaging [i.e. a positive diffusion-weighted imaging (DWI) abnormality].
2. Clinical syndrome not likely to represent transient ischemic attack (TIA) or other non-stroke etiology
3. Patient must be neurologically stable at the time of first MRI scan (i.e. stable NIH Stroke Scale score).
4. Initial MRI scan obtainable within 48 hours of symptom onset.
5. A pre-existing diagnosis of hypertension, either treated or untreated.
6. Average of two mean arterial blood pressures (separated by at least five minutes) at time of enrollment.

Exclusion Criteria:

1. Patients who have taken an angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) within seven (7) days of admission.
2. Patients who received intravenous or intra-arterial r-TPA for their current symptoms, or those who underwent mechanical thrombolysis.
3. Patients with hemorrhagic strokes, as seen on the initial head CT.
4. Patients with stroke-like symptoms, but no demonstrable lesion on DWI, or a DWI lesion < 2 cm in diameter (greatest dimension).
5. Patients with high-grade (>70%) internal carotid artery stenosis or occlusion ipsilateral to the current stroke.
6. Patients with high-grade aortic or mitral stenosis.
7. Patients with a previous adverse reaction to valsartan or other ARBs.
8. Patients with contraindications for MRI, including pacemakers, claustrophobia, or severe obesity.
9. Patients who are medically unstable for MR imaging, as determined by the treating team.
10. Patients with a severe co-existing disease that may interfere with the conduct of the study.
11. Patients receiving investigational drug therapies.
12. Informed consent cannot be obtained from the patient or an appropriate surrogate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08

PRIMARY OUTCOMES:
30 day glascow outcome score
30 day modified Rankin

CONTACTS AND LOCATIONS:
Overall Officials: Gregory W Albers, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States